CLINICAL TRIAL: NCT01946880
Title: An Investigator-Initiated, Phase II, Randomized, Withdrawal Study of Mycophenolate Mofetil (MMF) in Patients With Stable, Quiescent Systemic Lupus Erythematosus (SLE)
Brief Title: Randomized MMF Withdrawal in Systemic Lupus Erythematosus (SLE)
Acronym: ALE06
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ALE06; NIAID CRMS ID#: 20154 (Other: DAIT NIAID)
Record Dates: First submitted 2013-09-13; First posted 2013-09-20 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Systemic Lupus Erythematosus; SLE
Keywords: Systemic Lupus Erythematosus; Mycophenolate Mofetil (MMF)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Mycophenolic Acid; Hydroxychloroquine; Chloroquine; chloroquine diphosphate; Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate Mofetil Withdrawal (Experimental): These subjects will taper off MMF per the protocol-specified schedule over 12 weeks and remain off MMF for the rest of their study participation (up to Week 60 or until the primary endpoint of disease reactivation is met, whichever comes first).
  Interventions: Drug: Mycophenolate Mofetil; Drug: Hydroxychloroquine or Chloroquine; Drug: Prednisone
- Mycophenolate Mofetil Maintenance (Active Comparator): These subjects will continue MMF treatment (1000-3000 mg/day) for the rest of their study participation (up to Week 60).
  Interventions: Drug: Mycophenolate Mofetil; Drug: Hydroxychloroquine or Chloroquine; Drug: Prednisone

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Subjects will enter the trial on 1000-3000 mg/day of MMF and will be randomized to remain on MMF treatment or to be tapered off MMF within 12 weeks.
  Other Names: MMF
Drug: Hydroxychloroquine or Chloroquine — Subjects will be on concurrent anti-malarial agents (hydroxychloroquine or chloroquine). Hydroxychloroquine is approved by the FDA for the treatment of SLE. Hydroxychloroquine has been shown to help prevent flare in SLE, and to improve skin and musculoskeletal activity in particular.Even lupus nephritis outcomes appear improved on a background of hydroxychloroquine therapy
  Other Names: Plaquenil®; Chloroquine Phosphate®
Drug: Prednisone — Once the subject is randomized into the trial, the prednisone (or other corticosteroid) dose must be stable through Week 36 (24 weeks following protocol taper of MMF), in the absence of flares as described in Section 3.2 of the study protocol, Description of Primary Endpoint. Further taper of prednisone after that point is by the investigator's discretion based on the subject's clinical status.
  Other Names: corticosteroid

SUMMARY:
This trial seeks to describe the effect of withdrawal from mycophenolate mofetil (MMF) on risk of clinically significant disease reactivation in quiescent SLE patients who have been on long-term MMF therapy.

DETAILED DESCRIPTION:
Participants who have had inactive disease for at least 24 weeks will be enrolled. Half the subjects will continue on MMF and half the subjects will be tapered off their MMF within 12 weeks. All subjects will continue hydroxychloroquine and small doses of prednisone as needed. Subject visits to assess endpoints will occur every 4 weeks from Day 0 through Week 24 and then at Weeks 32, 40, 48, and 60.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent and comply with requirements of the study;
2. Age 18 - 70 years, inclusive, at randomization;
3. Diagnosis of SLE, per the American College of Rheumatology (ACR) criteria;
4. m-SLEDAI score < 4 at screening visit (SLEDAI score without serologies);
5. Physician Global Assessment (0-3) score of 1 or less at screening visit;
6. On a stable dose of MMF (1000-3000 mg/day) for at least 12 weeks prior to randomization;
7. Total duration of stable or decreasing MMF therapy must be at least:

   * two years for subjects initiating MMF for renal indications (with or without concurrent extra-renal manifestations), or
   * one year for subjects initiating MMF for extra-renal indications.
8. If the subject is on prednisone or other corticosteroid, the following criteria must be met:

   * the dose may not exceed 10 mg/day (or its equivalent) for the 12 weeks prior to randomization; however, temporary (up to 4 total days) increases, not to exceed 20mg/day, are permitted;
   * the dose must be held stable for the four weeks prior to randomization (no temporary increases within 4 weeks of randomization are permitted).
9. If the subject has a history of B cell depleting therapy within the past 3 years, presence of CD19 positive cells must be documented within 12 weeks prior to screening;
10. On maintenance HCQ or chloroquine at a stable dose for at least 12 weeks prior to randomization.

Exclusion Criteria:

1. A history of life-threatening neuropsychiatric SLE within 1 calendar year prior to randomization;
2. Any of the following laboratory abnormalities at the screening visit:

   * Proteinuria as defined by a spot protein/creatinine ratio > 1.0 mg/mg;
   * Serum creatinine > 2.0 mg/dL;
   * Transaminases > 2.5x the upper limit of normal (ULN);
   * Hemoglobin < 9 g/dL, unless the subject has documented hemoglobinopathy;
   * White blood count (WBC) < 2000/mm^3 (equivalent to < 2 x10^9/L);
   * Neutrophils < 1000/mm^3 (equivalent to < 1 x10^9/L); or
   * Platelet count < 75,000/mm^3 (equivalent to < 75 x 10^9/L).
3. Prednisone > 25 mg/day (or its equivalent) within 24 weeks prior to randomization for lupus activity;
4. Concomitant immunosuppressants including but not limited to azathioprine, methotrexate, 6-mercaptopurine, leflunomide, calcineurin inhibitors, anti-tumor necrosis factor agents within 12 weeks prior to randomization;
5. Plasmapheresis or IV immunoglobulin within 12 weeks prior to randomization;
6. Cyclophosphamide therapy within 24 weeks prior to randomization;
7. Concomitant therapy with belimumab within 24 weeks prior to randomization;
8. B cell depleting therapy within two calendar years of randomization;
9. Experimental therapy within the 24 weeks, or five half-lives of the agent, whichever is longer, prior to randomization;
10. Solid organ or stem cell transplantation;
11. Identified definitive diagnosis of another autoimmune disease that may require immunosuppression for treatment, including but not limited to: rheumatoid arthritis, scleroderma, primary Sjogren's syndrome, primary vasculitis, psoriasis, multiple sclerosis, ankylosing spondylitis, and inflammatory bowel disease.
12. Chronic infections including, but not limited to, human immunodeficiency virus (HIV), active tuberculosis (TB), currently receiving therapy)), hepatitis B or hepatitis C, or latent systemic fungal infection;
13. At or within 12 weeks of screening:

    * a history of or current positive purified protein derivative (PPD) (> 5 mm induration regardless of prior Bacillus Calmette-Guérin (BCG) vaccine administration) or positive QuantiFERON unless documentation exists of completion of at least one month of prophylaxis for latent TB or completed treatment for active TB; or
    * an indeterminate QuantiFERON® unless followed by a subsequent negative PPD or negative QuantiFERON.
14. History of malignancy within the last five years, except for resected basal or squamous cell carcinoma, treated cervical dysplasia, or treated in situ cervical cancer Grade I;
15. Pregnant or lactating, or intention to pursue pregnancy within three months after the completion of the study;
16. Unable or unwilling to use reliable methods of contraception, as outlined in the Mycophenolate REMS (e.g., Risk Evaluation and Mitigation Strategy), from four weeks prior to randomization to 6 weeks after completion of the study. This criterion applies to females of reproductive potential. (Reference: Mycophenolate REMS, Program Resources and Educational Materials, Information for Patients, What are my birth control options? Access the link at: (https://www.mycophenolaterems.com/PatientOverview.aspx).
17. Drug or alcohol abuse within one calendar year of randomization;
18. Other medical or psychiatric conditions that the investigator feels would place the subject at special risk by participation in this protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Chakravarty, MD, Study Chair — Oklahoma Medical Research Foundation; Judith A. James, MD, PhD, Study Chair — Oklahoma Medical Research Foundation
Locations (19):
- United States (19):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCSD, San Diego, California
  - UCSF School of Medicine, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Miami Hospitals and Clinics, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Feinstein Institute for Medical Research, Manhasset, New York
  - New York University, Langone Medical Center, New York, New York
  - Weill Cornell Medical College: Hospital for Special Surgery - Rheumatology Division, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Penn State University, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Chakravarty EF, Utset T, Kamen DL, Contreras G, McCune WJ, Aranow C, Kalunian K, Massarotti E, Clowse MEB, Rovin BH, Lim SS, Majithia V, Dall'Era M, Looney RJ, Erkan D, Saxena A, Olsen NJ, Ko K, Guthridge JM, Goldmuntz E, Springer J, D'Aveta C, Keyes-Elstein L, Barry B, Pinckney A, McNamara J, James JA. Mycophenolate mofetil withdrawal in patients with systemic lupus erythematosus: a multicentre, open-label, randomised controlled trial. Lancet Rheumatol. 2024 Mar;6(3):e168-e177. doi: 10.1016/S2665-9913(23)00320-X. Epub 2024 Jan 29. PMID 38301682
- [Derived] Wenderfer SE, Eldin KW. Lupus Nephritis. Pediatr Clin North Am. 2019 Feb;66(1):87-99. doi: 10.1016/j.pcl.2018.08.007. PMID 30454753
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nineteen study sites in the US were activated. A total of 123 participants were screened and 102 were randomized from November 2013 to May 2018.
Groups:
- MMF Maintenance: Participants received Mycophenolate Mofetil (MMF) treatment (1000-3000 mg/day) for the rest of their study participation (up to Week 60).
- MMF Withdrawal: Participants tapered off Mycophenolate Mofetil (MMF) per the protocol-specified schedule over 12 weeks and remained off MMF for the rest of their study participation (up to Week 60 or until the primary endpoint of disease reactivation was met, whichever came first).
Period: Overall Study
Arm/Group | MMF Maintenance | MMF Withdrawal
Started | 50 | 52
Completed | 43 | 49
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Met Primary Endpoint | 1 | 0
Not completed — Personal and Family Issues | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Maintenance: Participants received Mycophenolate Mofetil (MMF) treatment (1000-3000 mg/day) for the rest of their study participation (up to Week 60).
- Withdrawal: Participants tapered off Mycophenolate Mofetil (MMF) per the protocol-specified schedule over 12 weeks and remained off MMF for the rest of their study participation (up to Week 60 or until the primary endpoint of disease reactivation was met, whichever came first).
- Total: Total of all reporting groups
Arm/Group | Maintenance | Withdrawal | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 50 | 98
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.9) | 41.6 (12.5) | 42.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 47 | 86
  Male | 11 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 22
  Not Hispanic or Latino | 40 | 40 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 8 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 22 | 41
  White | 25 | 17 | 42
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 52 | 102
Disease Manifestation: Renal vs. Non-Renal Disease [Count of Participants; unit: Participants] — Renal disease, which included participants who had renal disease at screening as well as those who had renal manifestations in the past, versus non-renal disease, which included participants who never had renal disease.
  Participants
    Renal Disease | 40 | 38 | 78
    Non-Renal Disease | 10 | 14 | 24
Baseline MMF Dose [Count of Participants; unit: Participants] — Baseline dose of Mycophenolate Mofetil (MMF), defined as < 2000 mg per day versus ≥ 2000 mg per day.
  Participants
    < 2000 mg/day | 26 | 30 | 56
    ≥ 2000 mg/day | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Clinically Significant Disease Reactivation by Week 60
Description: Disease reactivation requires:1) SELENA-SLEDAI mild/moderate or severe flare,and 2) Increased immunosuppressive therapy on a sustained basis,defined by one of the following criteria:a) Sustained activity:Significant prolonged SLE flare requiring steroid increase/burst to ≥15 mg/day prednisone (or equivalent) for >4 weeks.b) Frequent relapsing/remitting:Participant flares requiring an increase/burst of steroids and is successfully tapered to <15 mg/day within 4 weeks, but this occurs on >2 occasions, or IA, IM or IV steroids on more than1 occasion.c)Clinical activity of sufficient severity to warrant resumption of/increased dose of MMF or addition of other major immunosuppressive including AZA or MTX.Regardless of steroid use, if the investigator observes disease activity of sufficient severity to warrant resumption, addition or increase in dosage of major immunosuppressant in the setting of a SELENA-SLEDAI flare, participant has met the primary endpoint.Risk difference also included
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The modified Intent-to-Treat (mITT) population included all randomized participants who begin ALE06-provided MMF and meet study entry criteria. Participants who, for whatever reason, do not complete their assigned therapy will be included in the mITT population in the groups to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 49 | 51
Participants | 5 | 9
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — The estimated risk difference (i.e. risk(MMF Withdrawal) - risk(MMF Maintenance)) and 95% confidence intervals around the risk difference at Week 60 were reported using the Kaplan-Meier product-limit estimator; Risk Difference (RD) = 0.07, 95% CI 2-sided [-0.068 to 0.214]

2. Secondary Outcome: Time to Clinically Significant Disease Reactivation
Description: The time to clinically significant disease reactivation was defined as the time from Baseline/Day 0 to the date of the first Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) assessment that met (or went on to meet) the criteria for clinically significant disease reactivation. Time to clinically significant disease reactivation was defined in study weeks as: date of SELENA-SLEDAI assessment that met reactivation criteria minus (-) baseline date.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The modified Intent-to-Treat (mITT) population included randomized participants who begin ALE06-provided MMF and meet study entry criteria. Participants who, for whatever reason, do not complete their assigned therapy will be included in the mITT population in the groups they were randomized. Participants who met disease reactivation were analyzed.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 5 | 9
Weeks | 38.0 (18.7) | 38.5 (19.6)

3. Secondary Outcome: Number of Participants Experiencing a Mild/Moderate or Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare by Week 60
Description: The SELENA-SLEDAI assesses systemic lupus erythematosus (SLE) disease activity and categorizes mild/moderate or severe flares based on changes in the SLEDAI score, the Physician's Global Assessment (PGA), medication use (prednisone, Nonsteroidal anti-inflammatory drugs, Plaquenil, major immunosuppressives), other disease activity criteria, and hospitalization due to SLE. An estimate of the risk difference ((i.e. risk(MMF Withdrawal) - risk(MMF Maintenance) and its corresponding 95% confidence interval (CI) were also included.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 49 | 51
Participants | 20 | 25
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other; Risk Difference (RD) = 0.08, 95% CI 2-sided [-0.116 to 0.279]

4. Secondary Outcome: Number of Participants Experiencing a Mild/Moderate or Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare by Week 60 Within the Lupus Nephritis Subgroup
Description: The SELENA-SLEDAI assesses systemic lupus erythematosus (SLE) disease activity and categorizes severe flares based on changes in the SLEDAI score, the Physician's Global Assessment (PGA), medication use (prednisone, Nonsteroidal anti-inflammatory drugs, Plaquenil, major immunosuppressives), other disease activity criteria, and hospitalization due to SLE. An estimate of the risk difference ((i.e. risk(MMF Withdrawal) - risk(MMF Maintenance) and its corresponding 95% confidence interval (CI) were also included.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The modified Intent-to-Treat (mITT) population included all randomized participants who begin ALE06-provided MMF and meet study entry criteria. Participants who, for whatever reason, do not complete their assigned therapy will be included in the mITT population in the group they were randomized. Participants in the renal subgroup were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 39 | 37
Participants | 15 | 19
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.13, 95% CI 2-sided [-0.091 to 0.360]

5. Secondary Outcome: Number of Participants Experiencing a Mild/Moderate or Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare by Week 60 Within the Non-Lupus Nephritis Subgroup
Description: as for outcome 4
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The modified Intent-to-Treat (mITT) population included all randomized participants who begin ALE06-provided MMF and meet study entry criteria. Participants who, for whatever reason, do not complete their assigned therapy will be included in the mITT population in the group they were randomized. Participants in the non-renal subgroup were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 10 | 14
Participants | 5 | 6
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.07, 95% CI 2-sided [-0.475 to 0.333]

6. Secondary Outcome: Number of Participants Experiencing a Mild/Moderate or Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare by Week 60 in the Baseline MMF<2000 mg/Day Subgroup
Description: The SELENA-SLEDAI assesses systemic lupus erythematosus (SLE) disease activity and categorizes severe flares based on changes in the SLEDAI score, the Physician's Global Assessment (PGA), medication use (prednisone, Nonsteroidal anti-inflammatory drugs, Plaquenil, major immunosuppressives), other disease activity criteria, and hospitalization due to SLE. An estimate of the risk difference ((i.e. risk(MMF Withdrawal) - risk(MMF Maintenance) and its corresponding 95% confidence interval (CI) were also included.
  MMF: mycophenolate mofetil
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The modified Intent-to-Treat (mITT) population included all randomized participants who begin ALE06-provided MMF and meet study entry criteria. Participants who, for whatever reason, do not complete their assigned therapy will be included in the mITT population in the group they were randomized. Baseline MMF <2000 mg/day participants were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 26 | 30
Participants | 11 | 13
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; The estimated risk difference (i.e. risk(MMF Withdrawal) - risk(MMF Maintenance)) and 95% confidence intervals around the risk difference at Week 60 were reported using the Kaplan-Meier product-limit estimator; Test type: Other; Risk Difference (RD) = -0.02, 95% CI 2-sided [-0.286 to 0.249]

7. Secondary Outcome: Number of Participants Experiencing a Mild/Moderate or Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare by Week 60 in the Baseline MMF ≥ 2000 mg/Day Subgroup
Description: as for outcome 6
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The modified Intent-to-Treat (mITT) population included all randomized participants who begin ALE06-provided MMF and meet study entry criteria. Participants who, for whatever reason, do not complete their assigned therapy will be included in the mITT population in the group they were randomized. Baseline MMF >=2000 mg/day participants were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 23 | 21
Participants | 9 | 12
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.20, 95% CI 2-sided [-0.090 to 0.497]

8. Secondary Outcome: Number of Participants Experiencing a Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare by Week 60
Description: as for outcome 4
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 49 | 51
Participants | 4 | 8
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.08, 95% CI 2-sided [-0.056 to 0.211]

9. Secondary Outcome: Number of Participants Experiencing a Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare by Week 60 Within the Lupus Nephritis Subgroup
Description: as for outcome 4
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 39 | 37
Participants | 3 | 7
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.12, 95% CI 2-sided [-0.041 to 0.284]

10. Secondary Outcome: Number of Participants Experiencing a Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare by Week 60 Within the Non-Lupus Nephritis Subgroup
Description: as for outcome 4
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 10 | 14
Participants | 1 | 1
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.04, 95% CI 2-sided [-0.285 to 0.206]

11. Secondary Outcome: Number of Participants Experiencing Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare by Week 60 in the Baseline MMF <2000 mg/Day Subgroup
Description: as for outcome 6
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 26 | 30
Participants | 3 | 6
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.09, 95% CI 2-sided [-0.118 to 0.289]

12. Secondary Outcome: Number of Participants Experiencing Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare by Week 60 in the Baseline MMF ≥ 2000 mg/Day Subgroup
Description: as for outcome 6
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 23 | 21
Participants | 1 | 2
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.05, 95% CI 2-sided [-0.103 to 0.212]

13. Secondary Outcome: Time to First Mild/Moderate or Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare
Description: The time to first mild/moderate or severe SELENA-SLEDAI flare was defined as the time from Baseline/Day 0 to the date of the first mild/moderate or severe SELENA-SLEDAI flare. Time to SELENA-SLEDAI flare was defined in study weeks as: date of SELENA-SLEDAI flare minus (-) baseline date. The SELENA-SLEDAI assesses systemic lupus erythematosus (SLE) disease activity and categorizes mild/moderate or severe flares based on changes in the SLEDAI score, the Physician's Global Assessment (PGA), medication use (prednisone, Nonsteroidal anti-inflammatory drugs, Plaquenil, major immunosuppressives), other disease activity criteria, and hospitalization due to SLE.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The modified Intent-to-Treat (mITT) population included randomized participants who begin ALE06-provided MMF and meet study entry criteria. Participants who, for whatever reason, do not complete their assigned therapy will be included in the mITT population in the groups they were randomized. Participants who had SELENA-SLEDAI flares were analyzed.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 20 | 25
Weeks | 20.5 (19.5) | 27.5 (16.7)

14. Secondary Outcome: Time to First Severe Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus-Disease Activity Index (SELENA-SLEDAI) Flare
Description: The time to first severe SELENA-SLEDAI flare was defined as the time from Baseline/Day 0 to the date of the first severe SELENA-SLEDAI flare. Time to severe SELENA-SLEDAI flare was defined in study weeks as: date of SELENA-SLEDAI flare minus (-) baseline date. The SELENA-SLEDAI assesses systemic lupus erythematosus (SLE) disease activity and categorizes mild/moderate or severe flares based on changes in the SLEDAI score, the Physician's Global Assessment (PGA), medication use (prednisone, Nonsteroidal anti-inflammatory drugs, Plaquenil, major immunosuppressives), other disease activity criteria, and hospitalization due to SLE.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 4 | 8
Weeks | 43.5 (9.9) | 41.5 (17.5)

15. Secondary Outcome: Number of Participants Experiencing Any British Isles Lupus Assessment Group (BILAG) A Flare by Week 60
Description: The BILAG assesses participants on a variety of disease activity criteria in nine body system categories (constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, ophthalmic, renal, and hematological). Each category is scored as an A, B, C, or D/E, where A indicates most severe disease activity and D/E indicates inactive/no disease activity. An estimate of the risk difference ((i.e. risk(MMF Withdrawal) - risk(MMF Maintenance) and its corresponding 95% confidence interval (CI) were also included.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 49 | 51
Participants | 1 | 4
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.06, 95% CI 2-sided [-0.028 to 0.149]

16. Secondary Outcome: Number of Participants in the Lupus Nephritis Subgroup Experiencing a British Isles Lupus Assessment Group (BILAG) A Renal Flare by Week 60
Description: as for outcome 15
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 39 | 37
Participants | 0 | 2
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.06, 95% CI 2-sided [-0.020 to 0.134]

17. Secondary Outcome: Change From Baseline in the Systemic Lupus International Collaborating Clinics/American College of Rheumatology Disease Damage Index for Systemic Lupus Erythematosus (SLICC/DI): Total Score
Description: The SLICC/DI measures accumulated damage that has occurred since the onset of systemic lupus erythematosus (SLE), regardless of cause, in 12 organ systems. SLE damage is defined as an irreversible change in an organ or system that has been present for at least 6 months. The SLICC/DI includes 39 areas of damage in 12 domains, where each item is rated as present or absent; if evidence of damage is present for a particular item, it is given a score of 1. Some items are scored with 2 or 3 points in the case of recurring events or end stage renal disease. The SLICC/DI total score will be computed as the sum of all scores for items indicated as present; scores can range from 0 to 45. Higher scores indicate more damage.
Time Frame: Baseline (Treatment Randomization) to Week 24, Week 48, and Week 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 49 | 51
Scores on a Scale
  Week 24 | 0.0 (0.15) | 0.0 (0.15)
  Week 48 | 0.0 (0.22) | 0.0 (0.15)
  Week 60 | 0.0 (0.37) | 0.0 (0.21)
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the SLICC/DI score between the treatment groups at Week 24; Test type: Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.1 to 0.1] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 24
Statistical Analysis 2: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the SLICC/DI score between the treatment groups at Week 48; Test type: Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.1 to 0.1] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 48
Statistical Analysis 3: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the SLICC/DI score between the treatment groups at Week 60; Test type: Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.1] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 60

18. Secondary Outcome: The Addition of Aggressive Adjunctive Therapy to Mycophenolate Mofetil (MMF) or Change in MMF Therapy to Cytotoxic Drug Due to Flare by Week 60
Description: The addition of aggressive adjunctive therapy could include intravenous (IV) immunoglobulin or rituximab at any point during the participant's study participation. A change in therapy to cytotoxic drug due to flare could include drugs such as cyclophosphamide, etc. A blinded list of study medications was reviewed to identify the addition of aggressive adjunctive therapy or cytotoxic drugs.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 49 | 51
Participants | 0 | 1
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.02, 95% CI 2-sided [-0.019 to 0.059]

19. Secondary Outcome: Cumulative Systemic Steroid Dose by Week 60
Description: Steroids include medications that code to a medication class which includes the terms "glucocorticoid" or "corticosteroid". Systemic steroids will include any of these steroids that are taken by mouth (PO), intravenous (IV), or intramuscular (IM). Total cumulative systemic steroid dose, in milligrams, was summarized over the 60 week study period, or until early study termination, for each participant.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: steroid dose (mg)
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 49 | 51
steroid dose (mg) | 851 (1148) | 912 (1995)

20. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy (FACIT-F) Fatigue Scale (FS): Total Score
Description: FACIT-Fatigue scale (FS) is a 13-item questionnaire completed by the patient (participant), that provides a measure of fatigue/quality of life, with a 7-day recall period. The participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-FS score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status. A decrease in the FACIT-FS score reflects worse fatigue/quality of life.
Time Frame: Baseline (Treatment Randomization) to Week 24, Week 48, and Week 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 49 | 51
units on a scale
  Week 24 | -2.41 (8.13) | -0.81 (10.62)
  Week 48 | -3.39 (7.53) | -0.85 (9.75)
  Week 60 | -3.13 (8.82) | 0.42 (9.05)
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the FACIT fatigue score between the treatment groups at Week 24; Test type: Other; Mean Difference (Final Values) = 1.61, 95% CI 2-sided [-2.24 to 5.45] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 24
Statistical Analysis 2: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the FACIT fatigue score between the treatment groups at Week 48; Test type: Other; Mean Difference (Final Values) = 2.54, 95% CI 2-sided [-1.13 to 6.21] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 48
Statistical Analysis 3: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the FACIT fatigue score between the treatment groups at Week 60; Test type: Other; Mean Difference (Final Values) = 3.55, 95% CI 2-sided [-0.17 to 7.28] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 60

21. Secondary Outcome: Change From Baseline in the Short Form Health Survey (SF-36) Physical Functioning (PF) Score
Description: The SF-36 is a 36-item, patient-reported survey of patient health. Higher scores indicate better outcomes while lower scores indicate more disability. The PF score is used to assess changes in physical functioning. It is scaled from 0 to 100 with a score of 0 equivalent to maximum disability and a score of 100 equivalent to no disability.
Time Frame: Baseline (Treatment Randomization) to Week 24, Week 48, and Week 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 49 | 51
Scores on a Scale
  Week 24 | -0.33 (4.05) | 0.22 (7.20)
  Week 48 | -0.49 (6.21) | 0.95 (6.13)
  Week 60 | -0.19 (5.63) | 1.79 (7.13)
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the PF score between the treatment groups at Week 24; Test type: Other; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-1.82 to 2.92] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 24
Statistical Analysis 2: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the PF score between the treatment groups at Week 48; Test type: Other; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [-1.14 to 4.03] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 48
Statistical Analysis 3: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the PF score between the treatment groups at Week 60; Test type: Other; Mean Difference (Final Values) = 1.98, 95% CI 2-sided [-0.71 to 4.67] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 60

22. Secondary Outcome: Change From Baseline in the Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score
Description: The SF-36 is a 36-item, patient-reported survey of patient health. Higher scores indicate better outcomes while lower scores indicate more disability. The Physical Component Score is comprised of the Physical Functioning Scale, the Role-Physical Scale, the Bodily Pain Scale, and the General Health Scale. It is scaled from 0 to 100 with a score of 0 equivalent to maximum disability and a score of 100 equivalent to no disability.
Time Frame: Baseline (Treatment Randomization) to Week 24, Week 48, and Week 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 49 | 51
Scores on a Scale
  Week 24 | -0.75 (4.82) | 0.90 (7.96)
  Week 48 | -1.92 (6.69) | 0.25 (6.83)
  Week 60 | -1.51 (6.66) | 1.51 (6.76)
Statistical Analysis 1: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the PCS score between the treatment groups at Week 24; Test type: Other; Mean Difference (Final Values) = 1.65, 95% CI 2-sided [-1.03 to 4.32] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 24
Statistical Analysis 2: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the PCS score between the treatment groups at Week 48; Test type: Other; Mean Difference (Final Values) = 2.17, 95% CI 2-sided [-0.69 to 5.02] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 48
Statistical Analysis 3: Comparison: MMF Maintenance vs MMF Withdrawal; Descriptive statistics (mean and 95% confidence interval) are reported for the difference in the change from baseline in the PCS score between the treatment groups at Week 60; Test type: Other; Mean Difference (Final Values) = 3.02, 95% CI 2-sided [0.22 to 5.82] — Estimate is for the difference in the change from baseline for MMF Withdrawal - MMF Maintenance at Week 60

23. Secondary Outcome: Change From Baseline in the Lupus Quality of Life (QoL)Score
Description: The Lupus QoL assessment is a 34 item questionnaire across 8 domains that is designed to find out how systemic lupus erythematosus (SLE) affects a participant's life over the preceding 4 weeks. Scores range from 0 (worst QoL) to 100 (best QoL). Domains include physical health, pain, planning, intimate relationships, burden to others, emotional health, body image, and fatigue.
Time Frame: Baseline (Treatment Randomization) to Week 24, Week 48, and Week 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 49 | 51
Scores on a Scale
  Change in Physical Health at Week 24 | -1.11 (9.20) | 1.04 (17.66)
  Change in Physical Health at Week 48 | -2.83 (11.57) | 0.46 (14.06)
  Change in Physical Health at Week 60 | 0.00 (9.02) | 1.56 (13.18)
  Change in Pain at Week 24 | -0.17 (10.67) | 1.77 (18.87)
  Change in Pain at Week 48 | -3.10 (12.73) | 1.60 (16.72)
  Change in Pain at Week 60 | -0.19 (12.39) | 1.42 (14.36)
  Change in Planning at Week 24 | 0.35 (16.75) | 3.90 (17.28)
  Change in Planning at Week 48 | -5.43 (16.66) | -0.18 (18.59)
  Change in Planning at Week 60 | -3.03 (16.48) | 0.18 (17.76)
  Change in Intimate Relationships at Week 24 | -1.47 (23.39) | 4.29 (18.68)
  Change in Intimate Relationships at Week 48 | -0.81 (10.67) | -1.10 (14.88)
  Change in Intimate Relationships at Week 60 | -2.08 (10.93) | 2.86 (13.92)
  Change in Burden to Others at Week 24 | 1.56 (21.99) | 0.18 (20.30)
  Change in Burden to Others at Week 48 | -0.58 (16.20) | -4.43 (16.56)
  Change in Burden to Others at Week 60 | -1.33 (17.14) | -3.55 (18.78)
  Change in Emotional Health at Week 24 | -0.87 (18.57) | 0.09 (13.02)
  Change in Emotional Health at Week 48 | -2.03 (15.71) | -1.22 (15.13)
  Change in Emotional Health at Week 60 | -1.52 (17.10) | -0.87 (13.06)
  Change in Body Image at Week 24 | 2.94 (16.12) | -1.09 (15.61)
  Change in Body Image at Week 48 | -0.17 (14.84) | -0.56 (17.76)
  Change in Body Image at Week 60 | 3.22 (15.29) | -4.45 (20.15)
  Change in Fatigue at Week 24 | 3.78 (16.04) | -1.17 (20.74)
  Change in Fatigue at Week 48 | -2.18 (18.04) | -1.56 (17.37)
  Change in Fatigue at Week 60 | -0.57 (15.36) | -1.95 (17.69)

24. Secondary Outcome: Time From Clinically Significant Disease Reactivation to Improvement in British Isles Lupus Assessment Group (BILAG) From Maximum Level During Flare
Description: For each participant who experienced disease reactivation, time from clinically significant disease reactivation to improvement in BILAG from maximum level (at least an A or B) during the flare was calculated in study days as: date of clinically significant disease reactivation minus (-) date of BILAG improvement. If multiple body systems had a BILAG flare at the visit, then the body system with the most severe score was tracked for improvement; if multiple body systems had the same score (at least an A or B), then just one needed to show improvement.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The modified Intent-to-Treat (mITT) population included all randomized participants who begin ALE06-provided MMF and meet study entry criteria. Participants who, for whatever reason, do not complete their assigned therapy will be included in the mITT population in the groups they were randomized. Participants who met primary endpoint were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 5 | 9
Days | 114.5 (123.7) | 40.5 (31.8)

25. Secondary Outcome: Time From Clinically Significant Disease Reactivation to Recovery to Baseline British Isles Lupus Assessment Group (BILAG) Score or BILAG C
Description: For each participant who experienced disease reactivation, time from clinically significant disease reactivation to recovery to baseline BILAG scores or BILAG C, whichever is worse, was calculated in study days as: date of clinically significant disease reactivation minus (-) date of BILAG recovery.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 5 | 9
Days | 114.5 (123.7) | 77.7 (63.4)

26. Secondary Outcome: Cumulative Excess Systemic Steroid Dose From Time of Clinically Significant Disease Reactivation to Return to Pre-Flare Dose or End of Trial Participation
Description: For each participant who experienced disease reactivation, excess systemic steroid dose was summed from the time of clinically significant disease reactivation until the dose returns to pre-flare levels or the end of study participation, whichever occurred first. Excess systemic steroid dose was defined as the total dose given for the flare minus (-) a participant's pre-flare steroid dose. Participants who do not have an increase in their steroid use due to the flare had their excess dose set to zero. Steroids include medications that code to a medication class which includes the terms "glucocorticoid" or "corticosteroid". Systemic steroids will include any of these steroids that are taken by mouth (PO), intravenous (IV), or intramuscular (IM).
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Steroid dose (mg)
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 5 | 9
Steroid dose (mg) | 812.8 (561.6) | 1750.7 (3384.6)

27. Secondary Outcome: Time From Clinically Significant Disease Reactivation to Return to Pre-Flare Steroid Dose
Description: For each participant who experienced disease reactivation, time from clinically significant disease reactivation to recovery to pre-flare steroid dose was calculated in study days as: date of clinically significant disease reactivation minus (-) date of return to pre-flare steroid dose.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 5 | 9
Days | NA (NA) — Six of the 14 subjects who met disease reactivation were on baseline steroids. Only 1 recovered to their baseline steroid dose. | 37 (NA) — Six of the 14 subjects who met disease reactivation were on baseline steroids. Only 1 recovered to their baseline steroid dose.

28. Secondary Outcome: Number of Grade 3, 4, or 5 Adverse Events (AEs) Related to Systemic Lupus Erythematosus (SLE)
Description: The number of Grade 3, 4, or 5 AEs classified as possibly, probably, or definitely related to SLE. The severity of AEs was classified using the National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The safety population (SP) includes all participants for whom study intervention was initiated.
Measure: Number; unit: Adverse Events
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 50 | 52
Adverse Events
  Grade 3 | 6 | 5
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

29. Secondary Outcome: Number of Grade 3, 4, or 5 Adverse Events (AEs) Related to Mycophenolate Mofetil (MMF)
Description: The number of Grade 3, 4, or 5 AEs classified as possibly, probably, or definitely related to MMF. The severity of AEs was classified using the National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The safety population (SP) includes all participants for whom study intervention was initiated.
Measure: Number; unit: Adverse Events
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 50 | 52
Adverse Events
  Grade 3 | 7 | 1
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

30. Secondary Outcome: Number of Grade 3, 4, or 5 Adverse Events (AEs)
Description: The number of Grade 3, 4, or 5 AEs. The severity of AEs was classified using the National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The safety population (SP) includes all participants for whom study intervention was initiated.
Measure: Number; unit: Adverse Events
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 50 | 52
Adverse Events
  Grade 3 | 18 | 15
  Grade 4 | 2 | 0
  Grade 5 | 0 | 0

31. Secondary Outcome: Number of Serious Adverse Events (SAEs).
Description: The number of SAEs. The severity of AEs was classified using the National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The safety population (SP) includes all participants for whom study intervention was initiated.
Measure: Number; unit: Serious Adverse Events
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 50 | 52
Serious Adverse Events | 12 | 6

32. Secondary Outcome: Number of Infection-Related Adverse Events (AEs)
Description: The number of AEs classified as infections. The severity of AEs was classified using the National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The safety population (SP) includes all participants for whom study intervention was initiated.
Measure: Number; unit: Adverse Events
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 50 | 52
Adverse Events | 63 | 49

33. Secondary Outcome: Number of Malignancies Reported as Adverse Events (AEs).
Description: The number of malignancies reported as AEs. The severity of AEs was classified using the National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The safety population (SP) includes all participants for whom study intervention was initiated.
Measure: Number; unit: Adverse Events
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 50 | 52
Adverse Events | 2 | 3

34. Secondary Outcome: Number of Grade 3, 4, or 5 Hematological Adverse Events (AEs).
Description: The number of Grade 3, 4, or 5 hematological AEs. The severity of AEs was classified using the National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The safety population (SP) includes all participants for whom study intervention was initiated.
Measure: Number; unit: Adverse Events
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 50 | 52
Adverse Events
  Grade 3 | 3 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

35. Secondary Outcome: Mortality Related to Systemic Lupus Erythematosus (SLE)
Description: Mortality related to SLE is defined as any death possibly, probably, or definitely related to SLE. The severity of AEs was classified using the National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The safety population (SP) includes all participants for whom study intervention was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 50 | 52
Participants | 0 | 0

36. Secondary Outcome: All-Cause Mortality
Description: All-cause mortality is defined as death from any cause occurring after randomization. The severity of AEs was classified using the National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Baseline (Treatment Randomization) to Week 60
Population: The safety population (SP) includes all participants for whom study intervention was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | MMF Maintenance | MMF Withdrawal
Number analyzed (Participants) | 50 | 52
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 weeks
Arm/Group | Maintenance | Withdrawal
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 7/50 | 5/52
Other Adverse Events (participants affected / at risk) | 38/50 | 41/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance (N=50) | Withdrawal (N=52)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 3 (3)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance (N=50) | Withdrawal (N=52)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 11 (17) | 13 (17)
Lymphopenia (Blood and lymphatic system disorders) | 8 (10) | 8 (9)
Neutropenia (Blood and lymphatic system disorders) | 5 (9) | 7 (9)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 2 (3) | 3 (3)
Tooth infection (Infections and infestations) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 14 (20) | 7 (11)
Urinary tract infection (Infections and infestations) | 6 (9) | 10 (11)
Blood creatinine increased (Investigations) | 3 (4) | 3 (5)
Glomerular filtration rate decreased (Investigations) | 6 (8) | 2 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (6) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Headache (Nervous system disorders) | 2 (3) | 5 (7)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 3 (6)

LIMITATIONS AND CAVEATS:
Enrollment ended early with 102 participants randomized instead of the planned 120.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT01946880/SAP_000.pdf
  • Study Protocol (2015-04-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT01946880/Prot_001.pdf